CLINICAL TRIAL: NCT06682676
Title: To Study the Diagnostic Efficacy of Cold Dry Air (CDA) Nasal Provocation Test in Patients With Idiopathic Rhinitis (IR)
Brief Title: Diagnostic Efficacy of CDA Nasal Provocation Test in Patients With IR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Cheng Lei, Professor， PhD, The First Affiliated Hospital with Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-SR-581
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic rhinitis (Experimental): Nasal ventilation tests were performed indoors at a temperature of (24±5) °C and a humidity of (70±10) %. Using acoustic rhinometry and rhinomanometry, total nasal volume, minimum cross-sectional area and total nasal resistance at 75Pa were recorded.Cold and dry air nasal provocation test usually requires nasal inhalation of 0°C-5°C, relative humidity < 10% cold air at a flow rate of 26L/min. The nasal symptom rating questionnaire and visual analogue scale were completed before and after the CDA test
  Interventions: Device: Nasal ventilation function test and cold and dry air nasal provocation test
- Healthy Volunteers (Experimental): Nasal ventilation tests were performed indoors at a temperature of (24±5) °C and a humidity of (70±10) %. Using acoustic rhinometry and rhinomanometry, total nasal volume, minimum cross-sectional area and total nasal resistance at 75Pa were recorded.Cold and dry air nasal provocation test usually requires nasal inhalation of 0°C-5°C, relative humidity < 10% cold air at a flow rate of 26L/min. The nasal symptom rating questionnaire and visual analogue scale were completed before and after the CDA test
  Interventions: Device: Nasal ventilation function test and cold and dry air nasal provocation test

INTERVENTIONS:
Device: Nasal ventilation function test and cold and dry air nasal provocation test — The visual analogue scale (VAS) of nasal symptoms, rhinoconjunctivitis quality of life questionnaire (RQLQ), total nasal symptom score (TNSS), total nasal volume (TNV), minimum cross-sectional area (MCA), peak inspiratory flow (PNIF), and total nasal resistance (TNR) at 75Pa were recorded before and after nasal ventilation function test and CDA nasal provocation test.

SUMMARY:
Chronic rhinitis is a common chronic nasal mucosal inflammatory disease. Its clinical symptoms and severity are diverse, mainly including allergic rhinitis, local allergic rhinitis, non-allergic rhinitis with hypereosinophilia syndrome and idiopathic rhinitis. All kinds of rhinitis have clinical symptoms such as nasal congestion, runny nose, sneezing, and nasal itching, but the causes are different. At present, the diagnosis of idiopathic rhinitis (IR) is based on detailed medical history and negative allergen test results, which is a diagnosis of exclusion. According to the position paper of the European Academy of Allergy and Clinical Immunology (EAACI), nasal hyperresponsiveness is an abnormal reaction of the nasal mucosa to stimuli that most people can tolerate. One of the distinguishing features of non-allergic rhinitis. cold dry air (CDA) nasal provocation test has been proved to be a good, safe and tolerable test for nasal hyperresponsiveness, with superior sensitivity and specificity. At present, there is still a lack of clear diagnostic criteria for IR. Therefore, optimizing CDA nasal provocation test, determining the diagnostic efficacy of CDA nasal provocation test with different parameters for IR, and initially constructing an IR diagnostic model can provide more comprehensive guidance for clinical diagnosis and treatment, which has important clinical significance.

DETAILED DESCRIPTION:
The visual analogue scale (VAS) of nasal symptoms, rhinoconjunctivitis quality of life questionnaire (RQLQ), total nasal symptom score (TNSS), total nasal volume (TNV), minimum cross-sectional area (MCA), peak inspiratory flow (PNIF), and total nasal resistance (TNR) at 75Pa were recorded before and after nasal ventilation function test and CDA nasal provocation test.

ELIGIBILITY:
Inclusion Criteria:

* IR patients: 1. Aged 18-65 years; 2. The presence of symptoms of rhinitis for more than 2 years, often triggered by non-specific stimuli, serum and nasal secretion allergen specific IgE test negative, nasal endoscopy examination ruled out severe anatomical disease and sinusitis with or without polyps, nasal secretion smear no eosinophils, allergic rhinitis, local allergic rhinitis, eosinophilia non-allergic rhinitis were excluded; 3. IR patients who visited the Department of Otorhinolaryngology, the First Affiliated Hospital of Nanjing Medical University and were willing to undergo CDA nasal provocation test; 4.Ptients who are willing to provide specimens for free to promote the study of the diagnostic efficacy of CDA nasal provocation test for IR.
* Healthy volunteers: 1. Aged 18-65 years; 2. Did not have any nasal symptoms and tested negative for allergens.

Exclusion Criteria:

* 1. Patients received glucocorticoids, immunomodulatory drugs, antihistamines, and other treatments that may affect the study results within the past 1 month. 2. Patients with unstable diseases (including severe asthma) and active immune system diseases; 3. Smoking; 4. Pregnant or lactating women; History of nasal surgery within 5.3 months; 6. Patients with any nasal conditions that may interfere with the efficacy or safety evaluation of CDA nasal provocation test; 7. Patients with low compliance and refusing to accept specimen and questionnaire collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-07 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire | 20min
  Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure
Visual Analog Score for pain | 20min
  Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure
Total nasal volume, minimum cross-sectional area, and total nasal resistance at 75Pa | 20min
  The total volume of nasal cavity, the minimum cross-sectional area and the total nasal resistance at 75Pa were recorded by acoustic rhinometer and rhinomanometer. The total nasal resistance was calculated by Rt=Rl*Rr/(Rl+Rr), Rt was the total nasal resistance, Rl and Rr represented the left and right nasal resistance respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Cheng, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No
All the individual participant data only available to reasearchers participated in this study